CLINICAL TRIAL: NCT00735475
Title: A Phase IV, Randomized, Observer-Blind, Multi-Center, Non Inferiority Comparison of the Immune Response of CSL Limited's Influenza Virus Vaccine Compared to a US Licensed Inactivated Split-Virion Influenza Vaccine in Adults Aged Greater Than or Equal to 65 Years
Brief Title: A Study to Determine the Immunogenicity and Safety Profile of CSL Limited's Influenza Virus Vaccine Compared to a US Licensed Comparator Influenza Virus Vaccine
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Seqirus (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: CSLCT-USF-07-41
Record Dates: First submitted 2008-08-13; First posted 2008-08-15 (Estimated); Results first posted 2011-09-01 (Estimated); Last update posted 2018-05-23 (Actual); Status verified 2018-04

CONDITIONS: Influenza
MeSH Terms: conditions — Influenza, Human | interventions — Afluria; Influenza Vaccines

STUDY DESIGN:
Who Masked: Investigator

ARMS (2):
- Afluria® (Experimental)
  Interventions: Biological: CSL Limited Influenza Virus Vaccine (Afluria®)
- Fluzone® (Active Comparator)
  Interventions: Biological: US Licensed Influenza Virus Vaccine (Fluzone®)

INTERVENTIONS:
Biological: CSL Limited Influenza Virus Vaccine (Afluria®) — A single 0.5 mL, intramuscular injection in the deltoid region of the arm on day 0.
  Arms: Afluria®
Biological: US Licensed Influenza Virus Vaccine (Fluzone®) — A single 0.5 mL, intramuscular injection in the deltoid region of the arm on day 0.
  Arms: Fluzone®

SUMMARY:
The purpose of this study is to determine the immunogenicity and safety profile of CSL Limited's Influenza Virus Vaccine compared to a US Licensed Comparator Influenza Virus Vaccine.

ELIGIBILITY:
Inclusion Criteria:

1. Males aged ≥ 65 years or females of non-childbearing potential aged ≥ 65 years ;
2. Written informed consent ;
3. Willingness to provide a blood sample.

Exclusion Criteria:

1. Known hypersensitivity to a previous dose of influenza vaccine or allergy to eggs, chicken protein, neomycin, polymyxin, or any components of the Study Vaccines;
2. Previous vaccination against influenza in 2008 or 2009 with seasonal trivalent inactivated influenza vaccine;
3. Known history of Guillain-Barré Syndrome;
4. Clinical signs of active infection and/or an oral temperature of greater than or equal to 100 degrees F (37.8 degrees C).
5. Have active or recent and clinically significant gastrointestinal/hepatic, renal, neurological, cardiovascular, respiratory, endocrine disorders or other medical disorders;
6. History of seizures;
7. Confirmed or suspected immunosuppressive condition, or a previously diagnosed immunodeficiency disorder;
8. Clinically significant history of malignancy
9. Current treatment, or treatment with radiotherapy or cytotoxic drugs at any time during the six months prior to administration of the Study Vaccine;
10. Current immunosuppressive or immunomodulative therapy;
11. Administration of immunoglobulins and/or any blood products within the 3 months preceding the administration of the Study Vaccine;
12. Participation in a clinical trial or use of an investigational compound within 30 days prior to receiving the Study Vaccine ;
13. Vaccination with a registered vaccine within 14 days (for inactivated vaccines) or 28 days (for live vaccines) prior to receiving the Study Vaccine.
14. Current treatment with warfarin or other anticoagulants;
15. Major congenital defects;
16. Evidence, or history (within the previous 12 months) of drug or alcohol abuse;
17. Unwillingness or inability to comply with the study protocol including completion of adverse event diary cards;
18. History of psychiatric disorders;
19. Resident of long term care facility.

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 1268 (Actual)
Dates: Start 2008-10; Primary Completion 2009-01 (Actual); Study Completion 2009-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Director Vaccines, Study Director — Seqirus
Locations (13):
- United States (13):
  - North Central Arkansas Medical Association, Mountain Home, Arkansas
  - Covance CRU, Inc, Boise, Idaho
  - The University of Iowa, Iowa City, Iowa
  - Kentucky Pediatric/ Adult Research, Bardstown, Kentucky
  - Saint Louis University Medical Center, St Louis, Missouri
  - University of Rochester School of Medicine and Dentistry, Rochester, New York
  - Duke University Medical Center, Durham, North Carolina
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Covance CRU, Inc., Portland, Oregon
  - Primary Physicians Research, Inc., Pittsburgh, Pennsylvania
  - Clinical Partners, LLC, Johnston, Rhode Island
  - Vanderbilt Medical Center, Nashville, Tennessee
  - Covance CRU Inc., Austin, Texas

RESULTS

PARTICIPANT FLOW:
Groups:
- Afluria® Group: Participants received one dose of the 2008/2009 formulation of Afluria® by intramuscular injection.
- Fluzone® Group: Participants received one dose of the 2008/2009 formulation of Fluzone® by intramuscular injection.
Period: Overall Study
Arm/Group | Afluria® Group | Fluzone® Group
Started | 631 | 637
Completed | 623 | 626
Not Completed | 8 | 11
Not completed — Adverse Event | 0 | 1
Not completed — Death | 1 | 1
Not completed — Lost to Follow-up | 3 | 3
Not completed — Physician Decision | 0 | 1
Not completed — Withdrawal by Subject | 4 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Afluria® Group | Fluzone® Group | Total
Number analyzed (Participants) | 630 | 636 | 1266
Age, Categorical [Count of Participants; unit: Participants] — Note: two participants (one in each group) did not provide follow-up safety information. Therefore, they are not included in the Safety Population.
  Participants
    <=18 years | 0 | 0 | 0
    Between 18 and 65 years | 0 | 0 | 0
    >=65 years | 630 | 636 | 1266
Age, Continuous [Mean (Standard Deviation); unit: years] | 71.7 (5.56) | 71.7 (5.53) | 71.7 (5.54)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 364 | 362 | 726
  Male | 266 | 274 | 540
Region of Enrollment [Number; unit: participants]
  United States | 630 | 636 | 1266

OUTCOME MEASURES:

1. Primary Outcome: Geometric Mean Titer 21 Days After the Study Vaccination
Time Frame: 21 days after vaccination
Population: Evaluable Population: comprised participants who were vaccinated, provided blood samples before and after vaccination, did not experience a laboratory-confirmed influenza infection, and did not receive a contraindicated medication.
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | Afluria® Group | Fluzone® Group
Number analyzed (Participants) | 622 | 630
Titers
  H1N1 (A/Brisbane/59/2007) | 58.60 [53.35 to 64.37] | 58.45 [53.23 to 64.17]
  H3N2 (A/Uruguay/716/2007) | 377.94 [339.31 to 420.97] | 337.23 [302.99 to 375.34]
  B (B/Florida/4/2006) | 30.16 [27.70 to 32.84] | 33.31 [30.54 to 36.33]

2. Primary Outcome: Percentage of Participants With Seroconversion 21 Days After the Study Vaccination
Description: Seroconversion rate was defined as the proportion of participants with a HI titer of less than 1:10 before vaccination achieving a HI antibody titer of 1:40 or more after vaccination, or with a HI titer of 1:10 or more before vaccination achieving a four-fold or greater increase in HI titer after vaccination.
Time Frame: 21 days after vaccination
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Afluria® Group | Fluzone® Group
Number analyzed (Participants) | 622 | 630
Percentage of participants
  H1N1 (A/Brisbane/59/2007) | 38.6 [34.7 to 42.5] | 43.2 [39.3 to 47.1]
  H3N2 (A/Uruguay/716/2007) | 69.0 [65.2 to 72.6] | 68.7 [64.9 to 72.3]
  B (B/Florida/4/2006) | 28.9 [25.4 to 32.7] | 33.8 [30.1 to 37.7]

3. Secondary Outcome: Frequency and Intensity of Local and Systemic Solicited Symptoms
Time Frame: 5 days after vaccination
Population: Safety Population: comprised all participants who received study vaccine and provided safety follow-up safety data.
Measure: Number; unit: Percentage of Participants
Arm/Group | Afluria® Group | Fluzone® Group
Number analyzed (Participants) | 630 | 636
Percentage of Participants
  Any local solicited symptom | 40.2 | 35.7
  Any tenderness | 36.2 | 31.4
  Any pain | 15.1 | 13.8
  Any swelling / induration | 7.1 | 7.9
  Any redness | 3.0 | 0.9
  Any bruising | 0.5 | 0.6
  Any systemic solicited symptom | 17.6 | 17.5
  Any headache | 8.6 | 10.5
  Any myalgia | 9.0 | 7.7
  Any malaise | 6.8 | 6.1
  Any chills | 2.2 | 2.4
  Any nausea | 1.7 | 1.4
  Any fever | 0.5 | 0.6
  Any vomiting | 0.3 | 0.3

4. Secondary Outcome: Duration of Local and Systemic Solicited Symptoms
Time Frame: 5 days after vaccination
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Afluria® Group | Fluzone® Group
Number analyzed (Participants) | 630 | 636
Days
  Any pain | 1.62 (2.094) | 1.70 (2.288)
  Any tenderness | 2.04 (2.147) | 1.90 (1.450)
  Any redness | 1.42 (0.692) | 2.67 (1.751)
  Any swelling / induration | 2.58 (3.031) | 2.25 (2.028)
  Any bruising | 6.50 (8.021) | 10.50 (9.883)
  Any fever | 1 (0) | 1 (0)
  Any headache | 2.08 (3.004) | 1.70 (1.782)
  Any malaise | 1.86 (1.850) | 2.08 (1.607)
  Any myalgia | 2.10 (3.193) | 2.65 (3.961)
  Any chills | 1.40 (0.737) | 2.29 (4.341)
  Any nausea | 1.62 (1.193) | 1.78 (0.972)
  Any vomiting | 1 (0) | 1 (0)

5. Secondary Outcome: Frequency and Intensity of Unsolicited Adverse Events (UAEs)
Description: Abbreviation UAE stands for Unsolicited Adverse Event.
Time Frame: 21 days after vaccination
Measure: Number; unit: participants
Arm/Group | Afluria® Group | Fluzone® Group
Number analyzed (Participants) | 630 | 636
participants
  Number of participants with at least one UAE | 169 | 171
  Number of participants reported Grade 1 UAE | 77 | 68
  Number of participants reported Grade 2 UAE | 57 | 68
  Number of participants reported Grade 3 UAE | 35 | 35

6. Secondary Outcome: Serious Adverse Events
Time Frame: 180 days after vaccination
Population: Safety Population: comprised all participants who received study vaccine and provided safety follow-up safety data.
Measure: Number; unit: participants
Arm/Group | Afluria® Group | Fluzone® Group
Number analyzed (Participants) | 630 | 636
participants
  Number of participants with at least one SAE | 22 | 26
  Number of participants with related SAE | 0 | 0

7. Secondary Outcome: New Onsets of Chronic Illness
Description: A NOCI was defined as the diagnosis of a chronic medical condition where the symptoms commenced or worsened following exposure to the study vaccine and may have included those potentially controllable by medication (e.g., glaucoma, hypertension).
Time Frame: 180 days after vaccination
Population: Safety Population: comprised all participants who received study vaccine and provided safety follow-up safety data.
Measure: Number; unit: participants
Arm/Group | Afluria® Group | Fluzone® Group
Number analyzed (Participants) | 630 | 636
participants
  Number of participants with at least one NOCI | 14 | 11
  Number of participants with related NOCI | 0 | 0
  Neoplasms benign, maligant and unspecified | 2 | 3
  Psychiatric disorders | 1 | 3
  Nervous system disorders | 0 | 1
  Eye disorders | 1 | 0
  Cardiac disorders | 2 | 0
  Vascular disorders | 3 | 1
  Gastrointestinal disorders | 1 | 1
  Hepatobiliary disorders | 1 | 0
  Musculoskeletal and connective tissue disorders | 2 | 2
  Renal and urinary disorders | 1 | 0
  Reproductive system and breast disorders | 2 | 0

ADVERSE EVENTS:
Time Frame: SAEs were collected up to 180 days after the study vaccination. Other adverse events were unsolicited adverse events that were collected up to 21 days after the study vaccination.
Description: Other Adverse Events reported were unsolicited adverse events that were collected up to 21 days after the study vaccination.
Arm/Group | Afluria® Group | Fluzone® Group
Serious Adverse Events (participants affected / at risk) | 22/630 | 26/636
Other Adverse Events (participants affected / at risk) | 142/630 | 119/636
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Afluria® Group (N=630) | Fluzone® Group (N=636)
Pneumonia (Infections and infestations) | 1 (1) | 2 (2)
Postoperative wound infection (Infections and infestations) | 1 (1) | 1 (1)
Diverticulitis (Infections and infestations) | 0 (0) | 1 (1)
Gastroenteritis (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia bacterial (Infections and infestations) | 1 (1) | 0 (0)
Tracheobronchitis (Infections and infestations) | 1 (1) | 0 (0)
Benign salivary gland neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Non-samall cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Non-small cell lung cancer stage IIIA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Intraventricular haemorrhage (Nervous system disorders) | 0 (0) | 1 (1)
Presyncope (Nervous system disorders) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 1 (1) | 0 (0)
Transient ischaemic attack (Nervous system disorders) | 0 (0) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Coronary artery disease (Cardiac disorders) | 4 (4) | 1 (1)
Acute myocardial infarction (Cardiac disorders) | 2 (2) | 2 (2)
Myocardial infarction (Cardiac disorders) | 0 (0) | 4 (4)
Atrial fibrillation (Cardiac disorders) | 3 (3) | 0 (0)
Cardiac failure congestive (Cardiac disorders) | 2 (3) | 0 (0)
Angina pectoris (Cardiac disorders) | 0 (0) | 2 (2)
Angina unstable (Cardiac disorders) | 2 (2) | 0 (0)
Bradycardia (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac arrest (Cardiac disorders) | 1 (1) | 0 (0)
Left ventricular dysfunction (Cardiac disorders) | 0 (0) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 1 (1) | 0 (0)
Hypertensive crisis (Vascular disorders) | 1 (1) | 0 (0)
Hypovolaemic shock (Vascular disorders) | 1 (1) | 0 (0)
Thrombophlebitis superficial (Vascular disorders) | 0 (0) | 1 (1)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Colitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Intervertebral disc degeneration (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Renal failure acute (Renal and urinary disorders) | 3 (3) | 0 (0)
Calculus baddder (Renal and urinary disorders) | 1 (1) | 0 (0)
Haematuria (Renal and urinary disorders) | 1 (1) | 0 (0)
Generalised oedema (General disorders) | 1 (1) | 0 (0)
Ankle fracture (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Anaemia postoperative (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Facial bones fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Femoral neck fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Hip fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Joint dislocation (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Postoperative ileus (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Pubic rami fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Therapeutic agent toxicity (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Afluria® Group (N=630) | Fluzone® Group (N=636)
Headache (Nervous system disorders) | 33 (43) | 22 (27)
Nasopharyngitis (Infections and infestations) | 9 (9) | 17 (18)
Sinusitis (Infections and infestations) | 5 (5) | 7 (7)
Upper respiratory tract infection (Infections and infestations) | 9 (9) | 3 (3)
Cough (Respiratory, thoracic and mediastinal disorders) | 8 (8) | 16 (16)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 14 (17) | 8 (8)
Rhinorrhea (Respiratory, thoracic and mediastinal disorders) | 11 (13) | 7 (7)
Myalgia (Musculoskeletal and connective tissue disorders) | 9 (10) | 8 (12)
Back pain (Musculoskeletal and connective tissue disorders) | 13 (16) | 3 (5)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 7 (10) | 9 (9)
Arthralgia (Musculoskeletal and connective tissue disorders) | 6 (9) | 8 (14)
Diarrhea (Gastrointestinal disorders) | 9 (10) | 8 (9)
Chills (General disorders) | 9 (10) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less